CLINICAL TRIAL: NCT04043806
Title: A Phase 3, Open-label Study Evaluating the Long-term Safety of VX-445 Combination Therapy in Subjects With Cystic Fibrosis
Brief Title: A Study Evaluating the Long-term Safety of VX-445 Combination Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX18-445-113; 2018-004652-38 (EudraCT Number)
Expanded Access: NCT04058210 (Approved for marketing)
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Results first posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ELX/TEZ/IVA (Experimental): Part A: Participants received ELX 200 milligram (mg) once daily (qd),TEZ 100 mg qd, and IVA 150 mg every 12 hours (q12h) in the treatment period for 96 weeks.
  Part B: Participants from certain countries participated in Part B and continued to received ELX 200 mg qd /TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 48 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed-dose combination (FDC) tablet for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
Drug: IVA — Tablet for oral administration.
  Other Names: VX-770; ivacaftor

SUMMARY:
This study evaluated the long-term safety and tolerability of elexacaftor (ELX), tezacaftor (TEZ), and ivacaftor (IVA) triple combination (TC) treatment in participants with cystic fibrosis (CF).

ELIGIBILITY:
Inclusion Criteria:

* Currently participating in study VX17-659-105 (NCT03447262)

Exclusion Criteria:

* History of drug intolerance in study VX17-659-105 that would pose an additional risk to the participant in the opinion of the investigator
* Current participation in an investigational drug trial (other than study VX17-659-105)

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (97):
- United States (46):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Miami Miller School of Medicine, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital Pulmonary and Sleep Medicine, Orlando, Florida
  - Johns Hopkins All Children's Hospital Outpatient Care Center, St. Petersburg, Florida
  - St. Luke's CF Center of Idaho, Boise, Idaho
  - Cystic Fibrosis Institute, Glenview, Illinois
  - Advocate Children's Hospital - Park Ridge / North Suburban Pulmonary and Critical Care Consultants, Niles, Illinois
  - Indiana University, Indianapolis, Indiana
  - The University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine / St. Louis Children's Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Albany Medical College, Pulmonary and Critical Care Medicine, Albany, New York
  - Lung and Cystic Fibrosis Center at Women and Children's Hospital of Buffalo, Buffalo, New York
  - Northwell Health- Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Santiago Reyes, M.D., Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Sanford Children's Speciality Clinic, Sioux Falls, South Dakota
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Children's Foundation Research Center / Le Bonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah / Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Pediatric Pulmonary & Cystic Fibrosis Clinic, Spokane, Washington
- Australia (7):
  - Royal Adelaide Hospital, Adelaide
  - The Prince Charles Hospital, Chermside
  - Alfred Hospital, Melbourne, VIC
  - Institute for Respiratory Health, Nedlands
  - Perth Children's Hospital, Nedlands
  - John Hunter Hospital & Hunter Medical Research Institute and John Hunter Children's Hospital, New Lambton
  - Queensland Children's Hospital, South Brisbane
- Canada (3):
  - Stollery Children's Hospital, Edmonton
  - Queen Elizabeth II Health Sciences Center, Halifax
  - St. Michael's Hospital, Toronto
- Juliane Marie Center, Rigshospitalet, Copenhagen, Denmark
- Germany (9):
  - Charite Paediatric Pulmonology Department, Berlin
  - Universitaetsklinkum Koeln, CF-Studienzentrum, Cologne
  - Ruhrlandklinik Westdeutsches Lungenzentrum am Klinikum Essen, Essen
  - Johann Wolfgang Goethe University, Frankfurt
  - Hannover Medical School, Hanover
  - Universitaetsklinikum Jena, Mukoviszidose-Zentrum, Jena
  - Universitatsklinikum Schleswig-Holstein, Klinik für Kinder- und Jugendmedizin, Lübeck
  - Klinikum Innenstadt, University of Munich, München
  - Pneumologisches Studienzentrum Muenchen-West, München
- Ireland (7):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Children's Health Ireland at Crumlin, Dublin
  - Children's Health Ireland at Temple Street, Dublin
  - St. Vincent's University Hospital, Dublin
  - University Hospital Galway, Galway
  - University Hospital Limerick (Adults), Limerick
- Israel (5):
  - Lady Davis Carmel Medical Center, Haifa
  - Pediatric Pulmonary Unit Rambam Medical Center, Haifa
  - Hadassah Medical Organization, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
  - Sheba Medical Center, Tel Litwinsky
- Klinika Mukowiscydozy IMD Oddozial Chorob Pluc Szpzoz IM. Dzieci WarszaWY, Łomianki, Poland
- Spain (7):
  - Hospital Universitari Vall d Hebron, Barcelona
  - Hospital Universitari Vall d´Hebron Servicio de Broncoscopia, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Infantil La Paz, Madrid
  - Parc Tauli Sabadell Hospital Universitari, Sabadell
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
- Switzerland (2):
  - Lindenhofspital - Quartier Bleu, Bern
  - Kinderspital Zuerich, Zurich
- United Kingdom (9):
  - Papworth Hospital NHS Foundation Trust, Papworth Everard, Cambridge
  - NHS Greater Glasgow and Clyde, Gartnavel General Hospital, Glasgow
  - St. James University Hospital, Leeds
  - Liverpool Heart and Chest Hospital, Liverpool
  - Royal Brompton & Harefield NHS Foundation Trust, Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, The Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Queens Medical Center, Nottingham
  - All Wales Adult Cystic Fibrosis Centre, University Hospital Llandough, Penarth

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent research/clinical-trial-data-sharing

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted as a single part study (Part A) in countries including United States (US) with commercially-available ELX/TEZ/IVA. The regional protocol for countries without commercially-available ELX/TEZ/IVA was amended so that participants in these countries had the opportunity to participate for up to an additional 48 weeks in Part B.
Pre-assignment Details: A total 458 participants were enrolled from the parent study VX17-659-105 (NCT03447262). One participant was enrolled but did not receive any dose in this study.
Period: Overall Study
Arm/Group | ELX/TEZ/IVA
Started | 458
Safety Set | 457 (Safety Set is defined as all participants who received at least 1 dose of study drug.)
Completed | 412
Not Completed | 46
Not completed — Commercial drug is available for participants | 13
Not completed — Physician Decision | 2
Not completed — Other | 12
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 6
Not completed — Other non-compliance | 2
Not completed — Withdrawal of Consent (not due to AE) | 8
Not completed — Never Dosed | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug were included in the baseline characteristics.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 457
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202
  Male | 255
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 437
  Not collected per local regulations | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 445
  Black or African American | 3
  Asian | 0
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0
  Not collected per local regulations | 5
  Multiple | 4

OUTCOME MEASURES:

1. Primary Outcome: Part A: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From Baseline through Week 100
Population: Safety set for included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- ELX/TEZ/IVA: Participants received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 96 weeks in Part A.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 457
participants
  Participants with TEAEs | 435
  Participants with SAEs | 75

ADVERSE EVENTS:
Time Frame: Day 1 Through Safety Follow-up Visit (up to Week 100 for Part A, up to Week 52 for Part B)
Description: The study was conducted as a single part study (Part A) in countries including United States (US) with commercially-available ELX/TEZ/IVA. The regional protocol for countries without commercially-available ELX/TEZ/IVA was amended so that participants in these countries had the opportunity to participate for up to an additional 48 weeks in Part B. The adverse events data has been reported for both the parts separately. MedDRA 25.0 applied for Part A and MedDRA 25.1 applied for Part B.
Groups:
- Part A: ELX/TEZ/IVA: Participants received ELX 200 mg qd, TEZ 100 mg qd, and IVA 150 mg q12h in the treatment period for 96 weeks.
- Part B: ELX/TEZ/IVA: Participants from certain countries participated in Part B and continued to received ELX 200 mg qd /TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 48 weeks.
Arm/Group | Part A: ELX/TEZ/IVA | Part B: ELX/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/457 | 0/66
Serious Adverse Events (participants affected / at risk) | 75/457 | 4/66
Other Adverse Events (participants affected / at risk) | 404/457 | 45/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: ELX/TEZ/IVA (N=457) | Part B: ELX/TEZ/IVA (N=66)
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 3 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Vascular device occlusion (General disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0
Herpes simplex pharyngitis (Infections and infestations) | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 31 | 1
Influenza (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 0
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 1 | 0
Stoma site discharge (Injury, poisoning and procedural complications) | 0 | 1
Human rhinovirus test positive (Investigations) | 0 | 1
Influenza A virus test positive (Investigations) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Piriformis syndrome (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Conversion disorder (Psychiatric disorders) | 1 | 0
Generalised anxiety disorder (Psychiatric disorders) | 1 | 0
Substance-induced mood disorder (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: ELX/TEZ/IVA (N=457) | Part B: ELX/TEZ/IVA (N=66)
Abdominal pain (Gastrointestinal disorders) | 30 | 2
Diarrhoea (Gastrointestinal disorders) | 33 | 1
Nausea (Gastrointestinal disorders) | 40 | 2
Vomiting (Gastrointestinal disorders) | 25 | 6
Fatigue (General disorders) | 46 | 4
Pain (General disorders) | 24 | 0
Pyrexia (General disorders) | 63 | 1
Immunisation reaction (Immune system disorders) | 42 | 1
COVID-19 (Infections and infestations) | 30 | 18
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 107 | 12
Nasopharyngitis (Infections and infestations) | 61 | 1
Sinusitis (Infections and infestations) | 31 | 3
Upper respiratory tract infection (Infections and infestations) | 71 | 10
Viral upper respiratory tract infection (Infections and infestations) | 46 | 0
Alanine aminotransferase increased (Investigations) | 39 | 3
Aspartate aminotransferase increased (Investigations) | 31 | 3
Blood creatine phosphokinase increased (Investigations) | 39 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 23 | 0
Headache (Nervous system disorders) | 92 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 114 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 41 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 52 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 61 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 27 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 24 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 36 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 26 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 67 | 0
Rash (Skin and subcutaneous tissue disorders) | 26 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT04043806/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT04043806/SAP_001.pdf